CLINICAL TRIAL: NCT00836784
Title: Comparing Efficacy of Old Versus New Toothbrushes in Plaque Removal in the Hands of 7-9 Year Old Children.
Brief Title: Comparison of New and 3-Month-Old Toothbrush in the Removal of Plaque in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Beheshte Malekafzali, Shahid beheshti medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 123456
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Plaque Removal
Keywords: Old tooth brush; Plaque removal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: old toothbrush
- 2 (Experimental)
  Interventions: Other: New tooth brush

INTERVENTIONS:
Other: old toothbrush — All children will receive new tooth brush 3 months before starting the study, at the end of 3 month the worn tooth brushes will be returned and the surface area within the outline will be determine using NIH (national institutes of health) image software.
  Other Names: worn toothbrush
  Arms: 1
Other: New tooth brush — The tooth brush which will be use in this study is "Jordan". A new Jordan toothbrush will be give to all children, and in "new tooth brush" group they will use these toothbrushes.
  Other Names: unused toothbrush
  Arms: 2

SUMMARY:
This study aimed to validate or invalidate non-inferiority in the plaque removal efficacy of old versus new toothbrushes in the hands of 7-9 year old children. This study was conducted in 93 Iranian students aged between 7-9 year old.

DETAILED DESCRIPTION:
At baselines, each student is given a new toothbrush which they will use for 3 months. The amount of wearing the 3-month-old brushes will determine by measurement of brushing surface areas using NIH imaging software. The outcomes will be measured after 3 month. The tooth brush which used in this study is "Jordan" with the following specifications: Length: 128 mm, 9 rows of bristles, 27 tufts, 24 monofilaments per tuft, height of monofilaments 10 mm and diameter of filaments 0.3 mm. The students will attend on two occasions following 48 hour periods of no oral hygiene. Following plaque scoring, students will brush with a new tooth brush at one visit and with a brush that they had used previously for 3 months at the other visit. Brushing time was 60 seconds. Plaque then will be re-scored and the percentage reduction in plaque score will be calculate using the Turesky plaque index. All plaque scoring will be performed by one examiner who is blind with the groups allocations.

ELIGIBILITY:
Inclusion Criteria:

1. subjects should be have central and lateral incisors, first permanent molar in each quadrant of maxilla and mandible
2. they should be without restoration on facial, lingual surfaces
3. subjects should be healthy without any disabilities

Exclusion Criteria:

1. subjects who wearing oral prosthesis,orthodontic brackets or removable appliances
2. subjects using mouthwashes which improve the oral hygiene

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Turesky plaque index | before and after brushing the teeth

CONTACTS AND LOCATIONS:
Overall Officials: Beheshte Malekafzali, Study Chair — Shahid Beheshti medical Science University; Mina Biria, Study Director — Shahid Beheshti medical Science University; Hoshyar Abbasi, Principal Investigator — Shahid Beheshti Medical Science University
Locations (1):
- Shahid Beheshti University, Tehran, Iran